CLINICAL TRIAL: NCT03546283
Title: Efficacy and Safety of Neuroprotectant Cattle Encephalon Glycoside and Ignotin Injection for Intracerebral Hemorrhage: a Multicenter, Randomized, Double-blinded, Placebo-controlled Trial.
Brief Title: Neuroprotectant for Hypertensive Intracerebral Hemorrhage
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rong Hu, MD (Other)
Responsible Party: Sponsor-Investigator, Rong Hu, MD, Director of neurosurgery, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neurosurg 04
Record Dates: First submitted 2018-05-16; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The patients with hypertensive intracerebral hemorrhage will be randomized into giving placebo group, the other treatments in this group follow the guidelines on the treatment of hypertensive intracerebral hemorrhage.
  Interventions: Drug: Placebos
- CEGI treatment (Experimental): The patients with hypertensive intracerebral hemorrhage will be randomized into giving drug CEGI, the other treatments in this group follow the guidelines on the treatment of hypertensive intracerebral hemorrhage.
  Interventions: Drug: Cattle Encephalon Glycoside and Ignotin

INTERVENTIONS:
Drug: Placebos — The patients with hypertensive intracerebral hemorrhage will be randomized into giving placebos, the other treatments in this group follow the guidelines on the treatment of hypertensive intracerebral hemorrhage.
  Arms: Control
Drug: Cattle Encephalon Glycoside and Ignotin — The patients with hypertensive intracerebral hemorrhage will be randomized into giving CEGI, the other treatments in this group follow the guidelines on the treatment of hypertensive intracerebral hemorrhage.
  Arms: CEGI treatment

SUMMARY:
Cattle encephalon glycoside and ignotin Cattle encephalon glycoside and ignotin (CEGI) injection (drug approval H22025046; Jilin Sihuan Pharmaceutical Co. LTD., Jilin, People's Republic of China) is a compound preparation of muscle extract from healthy rabbits and cattle brain gangliosides, which was approved by the Chinese Food and Drug Administration in 2011 and was commonly used as neuroprotectant in the treatment of central and peripheral nerve injuries in China. To evaluate the safety and efficacy of CEGI in treatment of Hypertensive intracerebral hemorrhage, we designed this study.

DETAILED DESCRIPTION:
Hypertensive intracerebral hemorrhage (HICH) is a type of stroke that is caused by hypertension-induced intracranial arterial, venous, and capillary ruptures. In recent years, the incidence of HICH has become higher, which has exposed society greatly to heavy social and economic burdens. Therefore it is necessary to find therapeutic strategies. ICH causes primary white matter injury by direct mechanical compression and hematoma expansion, and then it induces secondary injury through toxic product from the blood out of the vessel. The inﬂammatory response that follows ICH also contributes to the white matter injury. Additionally, post-ICH complications that include cortical thinning, cerebral edema, and hydrocephalus further aggravate the subcortical white matter damage.

The complex injury mechanisms that follow ICH implies that a multi-target neuroprotective agent might be able to achieve better neuroprotective eﬀects than current single-agent neuroprotective therapies.

Cattle encephalon glycoside and ignotin Cattle encephalon glycoside and ignotin (CEGI) injection (drug approval H22025046; Jilin Sihuan Pharmaceutical Co. LTD., Jilin, People's Republic of China) is a multi-target neuroprotective agent that includes polypeptides, various gangliosides, free amino acids and nucleic acids, which were extracted from muscle tissue of healthy rabbits and cattle brain gangliosides, and was approved by the Chinese Food and Drug Administration in 2011, commonly used as neuroprotectant in the treatment of central and peripheral nerve injuries in China.

It has been proven by basic research that CEGI treatment significantly alleviated the neurobehavioral dysfunction, promoted hematoma absorption, effectively up-regulated MBP/MAP-2 expression, and ameliorated white matter fiber damage [1]. CEGI was frequently used in the treatment of intracerebral hemorrhage, yet there is still a lack of high quality study to demonstrate its clinical efficacy. To achieve more clinical evidence of CEGI in treatment of Hypertensive intracerebral hemorrhage, we designed this study to further evaluate the efficacy and safety of CEGI in the treatment of Hypertensive intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18-75 years;
2. Newly diagnosed hypertensive intracerebral hemorrhage, bleeding position localizes in Basal ganglia and bleeding volume is within 25-50ml evaluated by head CT, and the hemorrhage does not break into lateral ventricle;
3. Obvious neurological dysfunction after onset, Glasco Comma Scale evaluation between 5-14, or NIHSS above 6, but without signs of cerebral hernia.
4. Enrolled within 72 hours after onset, and CT examination shows no hematomas expansion within 6 hours or above after diagnostic CT (hematoma expansion ≤ 5ml);
5. Written informed consent can be obtained.

Exclusion Criteria:

1. Diagnosed with intracerebral hemorrhage caused by aneurysm, brain tumor, trauma, cerebral parasitic disease, cerebrovascular malformation, moyamoya disease, cerebral arteritis, hematological diseases, or metabolic disorders;
2. Patients whose hematoma is unstable or progress leading to increased intracranial pressure;
3. Ever diagnosed with subarachnoid hemorrhage and ischemic stroke;
4. Ever received anticoagulants or antiplatelet drug treatment within one month prior to onset;
5. Abnormal coagulation function (platelet count <100×109/L, INR>1.4);
6. Patients who need operation treatment (including external ventricular drainage);
7. Patients who may suffer from mental or physical diseases that disturb outcome evaluation;
8. blood homocysteine higher than 15μmol/L when admission;
9. Patients who have serious diseases in heart, lung, liver, kidney, endocrine or hemopoietic system;
10. Allergic to protein or peptide;
11. Drug or alcohol addiction;
12. Pregnant women (positive in pregnancy test or lactating women)
13. Participated in other clinical trials within 3 months;
14. Patients considered as not suitable for clinical trials by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
GOSE at 90 days | 90 days after onset
  Glasgow Outcome Scale Extended at 90 days

SECONDARY OUTCOMES:
GOSE at 30 days | 30 days after onset
  Glasgow Outcome Scale Extended at 30 days
Score of mRS at 14days, 30 days and 90 days | 14 days, 30 days and 90 days after onset
  Global functional performance after stroke in terms of mRS at 14 days, 30 Days and 90 Days, respectively: 0 - No symptoms.1- No significant disability. Able to carry out all usual activities, despite some symptoms.2- Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.3- Moderate disability. Requires some help, but able to walk unassisted.4- Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.5- Severe disability. Requires constant nursing care and attention, bedridden, incontinent.6- Dead.
Score of NIHSS at 14days, 30 days and 90 days | 14 days, 30 days and 90 days after onset
  Global functional performance after stroke in terms of NIH Stroke Scale at 14 Days, 30 Days, and 90 Days, respectively: (0 = best possible, highest number = best possible) in areas of motor control of the arm (0-4), leg (0-4) sensory perception (0-2), language (0-3), limb ataxia (0-2), gaze (0-2), level of consciousness (0-3), level of consciousness -orientation (0-2), level of consciousness -commands (0-2), facial palsy (0-3), visual (0-3), dysarthria (0-2), and extinction (0-2).
Score of Barthel Index at 14days, 30 days and 90 days | 14 days, 30 days and 90 days after onset
  Global functional performance after stroke in terms of Barthel Index (scores 0~100) at 14 Days, 30 Days, and 90 Days, respectively: scores 100 mean good daily living ability; scores above 60 mean mild function disability that can live independently most time; scores between 60~41 mean moderate function disability that need some help in daily life; scores below 20 mean total disability that live helplessly.
Complications | within 90 days after onset
  Complications incidence including epilepsy, hydrocephalus, cerebral infarction, blooding recurrence, pneumonia and gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery , Southwest Hospital, Third Military Medical University,, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided